CLINICAL TRIAL: NCT06321510
Title: Real-World Treatment Patterns and Clinical Effectiveness of Dacomitinib in Advanced Non-Small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor-Positive in Taiwan
Brief Title: A Study to Learn About Dacomitinib in Patients With Non-small Cell Lung Cancer.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A7471070; NCT06321510 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: EGFR; NSCLC; brain; CNS; dacomitinib
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn about dacomitinib for the possible treatment of lung cancer.

This study is seeking participants who:

* have lung cancer that could not be controlled.
* have a type of gene called epidermoid growth factor receptor. A gene is a part of your DNA that has instructions for making things your body needs to work.
* have received dacomitinib for their lung cancer.

All participants in this study had received dacomitinib. Dacomitinib is a tablet that is taken by mouth at home. They continued to take dacomitnib until their cancer was no longer responding. The study will look at the experiences of people receiving the study medicine. This will help to see if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of histologically or cytologically confirmed diagnosis of advanced NSCLC with EGFR-activating mutations detected by an appropriate test
* Patients who were treated with dacomitinib as first-line treatment for advanced NSCLC during 01 October 2020 to 31 December 2022.
* Age ≥18 years old
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients who have been treated with any systemic anti-cancer therapies within 12 months prior to dacomitinib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer and treated with dacomitnib in medical center or regional hospital will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with dacomitinib dosage change and reasons | 52 months from index date
  The percentage of patients with dacomitinib dosage change and reason during follow-up period will be summarized.
Percentage of patients with dacomitinib treatment discontinuation | 52 months from index date
  The percentage of patients with dacomitinib treatment discontinuation for any reason during follow-up period will be summarized.

SECONDARY OUTCOMES:
Real-world overall survival (rwOS) | 52 months from index date
  Time to death from index date during follow-up period will be summarized by K-M plot with corresponding 95% CI.
Real-world progression-free survival | 52 month from index date
  Time to real-world disease progression or death, which ever occurs first, during follow-up period will be summarized by K-M plot with corrsponding 95% CI.
Real-world best objective response rate (rwORR) | 52 months from index date
  Number and percentage of patients achieving real-worl overall response (CR or PR).
real-world intracranial response rate (rwIC-ORR) | 52 months from index date
  The percentage of patients achieving real-world intracranial response (CR or PR) for brain metastases during follow-up period will be summarized.
real-world extracranial response rate (rwEC-ORR) | 52 months from index date
  The percentage of patients achieving real-world extracranial response (CR or PR) for brain metastases during follow-up period will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A7471070